CLINICAL TRIAL: NCT00000313
Title: Predictive Values of Serotonergic Alterations for Outcome
Brief Title: Predictive Values of Serotonergic Alterations for Outcome - 2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: NIDA-09468-2; R01-09468-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2002-12

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Fenfluramine

INTERVENTIONS:
Drug: Fenfluramine

SUMMARY:
The purpose of this study is to evaluate the predictive value of serotonergic alterations for outcome.

ELIGIBILITY:
Please contact site for information.

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0

PRIMARY OUTCOMES:
Side effects
Neuroendocrine changes
Psychological changes
Craving

CONTACTS AND LOCATIONS:
Overall Officials: Laure Buydens-Branchey, M.D., Principal Investigator — VA Medical Center
Locations (1):
- VA Medical Center, Brooklyn, New York, United States